CLINICAL TRIAL: NCT02708615
Title: A Randomized Controlled Trial of Gynecological Speculum Examination: Straight Horizontal Insertion vs. Vertical Insertion and Rotation
Brief Title: Gynaecological Speculum Examination: Straight Horizontal Insertion Versus Vertical Insertion and Rotation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15-082
Record Dates: First submitted 2016-03-02; First posted 2016-03-15 (Estimated); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Vaginal Speculum Examination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vertical rotation (Other): Vertical insertion and 90 degree rotation of speculum in vagina
  Interventions: Other: Type of speculum vaginal insertion method
- Straight horizontal insertion (Other): Straight horizontal insertion of speculum with no rotation in vagina
  Interventions: Other: Type of speculum vaginal insertion method

INTERVENTIONS:
Other: Type of speculum vaginal insertion method — Speculum insertion type will either be vertical rotation (as per common practice in Canada) or straight horizontal insertion

SUMMARY:
This study compares two different types of speculum insertion to determine the level of discomfort they might cause. This study compares the straight horizontal insertion (SHI) of the speculum and the vertical insertion and rotation (VIR).

Participants are randomly assigned to one of the two insertion groups and are not told which group they are in until the examination is over. Participants rate their level of discomfort immediately after insertion of the speculum.

Basic demographic information (e.g., age, ethnicity, number of vaginal deliveries, menopausal status, etc.) and clinical information are also collected to determine if other factors influence the level of discomfort experienced.

*NOTE* This is NOT a paid study.

DETAILED DESCRIPTION:
In most medical schools around the world, speculum examination is taught using a bivalved speculum, since this is the type of speculum most commonly used in clinical practice. Due to the oval shape of the vulva, and the alignment of the labia majora and minora, the aperture of vaginal introitus is commonly perceived to have a vertical orientation. In reality however, the vaginal introitus is round and the vagina itself has more of a horizontal orientation: the anterior and posterior vaginal walls are opposed, and the sidewalls only become apparent once the anterior and posterior walls are separated. Nevertheless, the most common way of teaching the speculum examination worldwide is to introduce the speculum in a vertical orientation and then once it is successfully inserted into the vagina to rotate it 90° into a horizontal position. Once it is correctly positioned, it is slowly opened to visualize the vaginal epithelium and the cervix. However, in clinical practice, the rotation of the speculum in the vagina may cause pain and discomfort. Introduction of the speculum initially in a horizontal orientation, without rotation in the vagina, seems more appropriate and could potentially be associated with less discomfort or pain for women undergoing this exam. In practice, a minority of clinicians separate the labia first, introduce the speculum in a direct horizontal fashion, and thus avoid the potentially uncomfortable twisting part of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 18 years of age or older
* Undergoing a speculum examination as part of their regular clinical care
* Proficient knowledge of the English language and able to sign the informed consent form

Exclusion Criteria:

* Younger than 18 years of age
* Women with a history of vulvodynia, vaginismus, or dyspareunia
* No prior sexual activity or intercourse
* Active vaginal, cervical, uterine or adnexal infection
* Active pregnancy or within 6 weeks postpartum
* Vulvar or vaginal surgery within three months
* Psychiatric conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-11-27 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2021-11-27 (Actual)

PRIMARY OUTCOMES:
Pain/discomfort ratings of women receiving straight horizontal speculum insertion vs. those receiving vertical speculum insertion and rotation, as measured by a visual analog scale | Measured immediately after speculum insertion
  The primary objective of this study is to quantify the amount of pain/discomfort women experience with two different types of speculum insertion: straight horizontal insertion (SHI) and vertical insertion and rotation (VIR). Participants will rate their pain/discomfort by placing a mark on a visual analog scale measuring 10 cm in length. Pain/discomfort ratings on this scale range from "no pain" to "pain as bad as it possibly could be".

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yudin, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No